CLINICAL TRIAL: NCT03986710
Title: Feasibility and Performance of a Novel 3D Virtual Treatment Planning Software: Single Surgeon Study
Acronym: IPSCD-TIM-GS
Status: Completed | Type: Observational
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Gwen Swennen, maxillofacial surgeon, principal investigator, AZ Sint-Jan AV
Other Study IDs: 2004
Record Dates: First submitted 2019-02-14; First posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Orthognathic Surgery
Keywords: 3D virtual planning software; timing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background Three-dimensional (3D) imaging and subsequent 3D virtual treatment planning are becoming state of the art in orthognathic surgery. However, current available software is still too time-consuming. KLS Martin (Tuttlingen, Germany) has currently completed the preclinical phase of their novel 3D virtual planning software, "IPS (Individual Patient Solutions) CaseDesigner (IPSCD)".

Objectives The authors aim to test pre-release versions of the IPSCD software under real-world working conditions by a single surgeon.In specific, the authors aim to demonstrate that the IPSCD will ensure a significant reduction in treatment planning time.

Study design closed beta-phase Patients presenting at the division of maxillofacial surgery at the different hospital centers, for an orthognathic-related problem will receive a complete routine work-up, including a cone-beam CT (CBCT) according to the IPSCD protocol. The same surgeon will run all the virtual planning steps with both conventional software (Maxilim) and the novel software. Timing of the eight major steps will be measured with a digital chronometer.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all ages
* Patients of both genders
* Patients should present themselves at the division of Maxillofacial surgery
* Patients should receive standardized cone-beam computed tomography (CBCT) image acquisition, according to the IPSCD protocol
* Preoperative 3D virtual planning should be performed by the same surgeon

Exclusion Criteria:

* All patients that do not fit the abovementioned description
* Patients with posttraumatic deformity
* Patients with congenital deformity
* Patients with pre-prosthetic indication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: consecutive orthognathic patients operated and planned by a single surgeon (GS)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
duration of total 3D virtual treatment planning time | preoperative
  duration of total 3D virtual treatment planning time, measured in seconds with a digital online chronometer

SECONDARY OUTCOMES:
duration of 8 major steps in 3D virtual treatment planning | preoperative
  duration of 8 major steps in 3D virtual treatment planning, measured in seconds with a digital online chronometer

CONTACTS AND LOCATIONS:
Overall Officials: Gwen Swennen, Principal Investigator — AZ Sint-Lucas Brugge

IPD SHARING:
Plan to Share IPD: No